CLINICAL TRIAL: NCT03598608
Title: A Phase 1/Phase 2 Clinical Study to Evaluate the Safety and Efficacy of a Combination of MK-4280 and Pembrolizumab (MK-3475) in Participants With Hematologic Malignancies
Brief Title: Study to Evaluate the Safety and Efficacy of a Combination of Favezelimab (MK-4280) and Pembrolizumab (MK-3475) in Participants With Hematologic Malignancies (MK-4280-003)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4280-003; MK-4280-003 (Other: MSD); 2023-503587-17-00 (Registry Identifier: EU CT); U1111-1287-5405 (Registry Identifier: UTN); 2018-001461-16 (EudraCT Number)
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Masking Description: Participants in Part B: Randomized cHL-Monotherapy arm in the study will be randomized (1:1 ratio) to receive pembrolizumab or favezelimab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: Favezelimab Dose A+pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab by intravenous (IV) infusion followed by favezelimab Dose A by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab
- Part A: Favezelimab Dose B+pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab by IV infusion followed by favezelimab Dose B by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab
- Part A: Favezelimab Dose C+Pembrolizumab (Experimental): Participants receive 200 mg pembrolizumab by IV infusion followed by favezelimab Dose C by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab
- Part B: cHL-Combination Therapy (Experimental): Participants with cHL receive 200 mg pembrolizumab by IV infusion followed by the recommended Phase 2 dose (RP2D) of favezelimab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab
- Part B: DLBCL-Combination Therapy (Experimental): Participants with DLBCL receive 200 mg pembrolizumab by IV infusion followed by the RP2D of favezelimab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab
- Part B: iNHL-Combination Therapy (Experimental): Participants with iNHL receive 200 mg pembrolizumab by IV infusion followed by the RP2D of favezelimab by IV infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab
- Part B: Randomized cHL-Monotherapy (Experimental): Participants with cHL receive either pembrolizumab by IV infusion or the RP2D of favezelimab by IV infusion on Day 1 of each 3-week cycle (Q3W) for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: pembrolizumab; Biological: Favezelimab

INTERVENTIONS:
Biological: pembrolizumab — Administered as an IV infusion every 3 weeks (Q3W)
  Other Names: KEYTRUDA®; MK-3475
Biological: Favezelimab — Administered as an IV infusion Q3W
  Other Names: MK-4280

SUMMARY:
This study will evaluate the safety and efficacy of favezelimab (MK-4280) in combination with pembrolizumab (MK-3475) using a non-randomized study design in participants with the following hematological malignancies:

* classical Hodgkin lymphoma (cHL)
* diffuse large B-cell lymphoma (DLBCL)
* indolent non-Hodgkin lymphoma (iNHL)

This study will also evaluate the safety and efficacy of pembrolizumab or favezelimab administered as monotherapy in participants with cHL using a 1:1 randomized study design.

The study will have 2 phases: a safety lead-in and an efficacy expansion phase. The recommended Phase 2 dose (RP2D) will be determined in the safety lead-in phase by evaluating dose-limiting toxicities.

There is no primary hypothesis for this study.

DETAILED DESCRIPTION:
Per protocol amendment 7, the secondary serum concentration endpoints were removed and will not be reported.

ELIGIBILITY:
Inclusion Criteria:

* Has measurable disease, defined as ≥1 lesion that can be accurately measured in 2 dimensions with diagnostic quality cross sectional anatomic imaging (computed tomography or magnetic resonance imaging). Minimum measurement must be >15 mm in the longest diameter or >10 mm in the short axis
* Is able to provide a core or excisional tumor biopsy for biomarker analysis from an archival (within 3 months) or newly obtained biopsy at screening
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG)

Exclusion Criteria:

* Has known clinically active central nervous system (CNS) involvement
* Has received prior therapy with an anti-lymphocyte activation gene-3 (LAG-3) antibody
* Has received chimeric antigen receptors (CAR)-T-cell therapy for cHL and DLBCL Cohorts
* Has received prior anticancer therapy or thoracic radiation therapy within 14 days before the first dose of study treatment
* Has ≥Grade 2 non-hematological residual toxicities from prior therapy
* Has had a prior anticancer monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤Grade 1 or at baseline) from AEs due to agents administered ≥4 weeks earlier
* Has received a live vaccine within 30 days prior to first dose of study treatment. Administration of killed vaccines are allowed
* Has received an investigational agent or used an investigational device within 4 weeks prior to intervention administration
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Has a known additional malignancy that is progressing or requires active treatment with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has an active infection requiring intravenous systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has known, active hepatitis B or hepatitis C infection
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has had an allogeneic hematopoetic stem cell/solid organ transplantation within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing a Dose-limiting Toxicity (DLT) | Cycle 1 (up to 21 days)
  DLT will be defined as any drug-related adverse event (AE) observed during the DLT evaluation period (Cycle 1) that results in a change to a given dose or a delay in initiating the next cycle and reported as the percentage of participants experiencing a DLT defined by the National Cancer Institute Common Terminology for Adverse Events version 4.0.
Percentage of Participants Experiencing an Adverse Event (AE) | From time of signing informed consent form (ICF) until the end of follow-up (up to approximately 27 months)
  Percentage of participants experiencing an AE defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study treatment
Percentage of Participants with Treatment Discontinuations Due to an AE | From time of signing informed consent form (ICF) until the end of study treatment (up to approximately 24 months)
  Percentage of participants discontinuing study treatment due to an AE

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants in the analysis population who had a Complete Response or a Partial Response per lymphoma disease response criteria (Cheson et. al., 2007) as assessed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (25):
- United States (8):
  - Banner MD Anderson Cancer Center ( Site 0020), Gilbert, Arizona
  - City of Hope ( Site 0001), Duarte, California
  - Ronald Reagan UCLA Medical Center (Radiological Sciences) ( Site 0007), Los Angeles, California
  - Pacific Cancer Care ( Site 0006), Monterey, California
  - University of California San Francisco ( Site 0023), San Francisco, California
  - Dana Farber Cancer Institute ( Site 0002), Boston, Massachusetts
  - Fox Chase Cancer Center ( Site 0019), Philadelphia, Pennsylvania
  - Texas Oncology-Austin Midtown ( Site 8002), Austin, Texas
- Australia (4):
  - Concord Repatriation & General Hospital ( Site 0203), Concord, New South Wales
  - Princess Alexandra Hospital ( Site 0204), Woollongabba, Queensland
  - Monash Health ( Site 0201), Clayton, Victoria
  - St Vincent s Hospital (Melbourne) Limited ( Site 0202), Fitzroy, Victoria
- Canada (4):
  - BC Cancer ( Site 0107), Vancouver, British Columbia
  - CancerCare Manitoba ( Site 0101), Winnipeg, Manitoba
  - Princess Margaret Cancer Centre ( Site 0100), Toronto, Ontario
  - Jewish General Hospital ( Site 0105), Montreal, Quebec
- Germany (2):
  - U. klinikum Koeln AOER ( Site 0326), Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig AOeR ( Site 0327), Leipzig, Saxony
- Israel (4):
  - Rambam Medical Center ( Site 0382), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 0383), Jerusalem
  - Chaim Sheba Medical Center. ( Site 0380), Ramat Gan
  - Sourasky Medical Center ( Site 0381), Tel Aviv
- Italy (3):
  - A.O. Universitaria Policlinico S. Orsola-Malpighi ( Site 0351), Bologna, Emilia-Romagna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori ( Site 0354), Meldola, Forli-Cesena
  - Humanitas-U.O di Oncologia medica ed Ematologia ( Site 0352), Rozzano, Milano

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Derived] Armand P, Zinzani PL, Timmerman J, Johnson NA, Lavie D, Thiagarajan K, Topp BG, Pillai P, Herrera AF. Estimating efficacy of favezelimab plus pembrolizumab relative to pembrolizumab in anti-PD-1-refractory Hodgkin lymphoma. Blood Adv. 2025 Oct 14;9(19):4987-4995. doi: 10.1182/bloodadvances.2024014654. PMID 40668662
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26283&tenant=MT_MSD_9011